CLINICAL TRIAL: NCT01609439
Title: Pre-operative Vitamin D Supplementation to Reduce Post-operative Hypocalcemia in Patients Undergoing Total Thyroidectomy: A Randomized Controlled Trial
Brief Title: Preoperative Vitamin D for Post-thyroidectomy Hypocalcemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Caroline Xu, Resident, Otolaryngology-Head and Neck Surgery, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: UAH-Oto-TT01
Record Dates: First submitted 2012-05-24; First posted 2012-06-01 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2012-05

CONDITIONS: Hypocalcemia
Keywords: Permanent; temporary; hypocalcemia
MeSH Terms: conditions — Hypocalcemia | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment (Experimental): Pre-operative Vitamin D 800 units x 4 weeks
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 800 units for 4 weeks preoperatively
  Arms: Treatment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if pre-operative vitamin D supplementation lowers the incidence of post-operative transient or permanent hypoparathyroidism in patients undergoing total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total thyroidecomty +/- CND
* Adult (age > or = 18)

Exclusion Criteria:

* Known chronic kidney disease
* Known primary hyper or hypoparathyroidism
* Known hypoalbuminemia
* Concurrent use medications affecting calcium metabolism
* Completion hemithyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Hypocalcemia | Transient (<72 hrs post-operatively)
  Clinical signs and symptoms(paraesthesias, etc.) OR Laboratory evidence (ICa < 0.9) Need for IV calcium supplementation

SECONDARY OUTCOMES:
Hypocalcemia | Permanent (>4 weeks)
  ICa at 6 weeks and need for continued supplementation beyond 6 weeks post-op (i.e. 3 months follow-up post-operatively)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada